CLINICAL TRIAL: NCT00779428
Title: Phase 2 Clinical Trial of Tanespimycin in Patients With Advanced Malignancies After Failure of Previous Anti-cancer Therapy Regimens Who Have Participated on a Prior Protocol Investigating Tanespimycin
Brief Title: Clinical Trial of Continuing Treatment for Patients Who Have Participated on a Prior Protocol Investigating Tanespimycin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA200-002
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Malignancies
Keywords: This is an open-label continuing treatment protocol in patients with advanced malignancies who will receive Tanespimycin
MeSH Terms: interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Tanespimycin

INTERVENTIONS:
Drug: Tanespimycin — Solution, IV
  This is a one arm study with the dose, frequency, and duration assigned as per previous protocol (KOS-953, 17-AAG)
  Other Names: BMS-722782

SUMMARY:
The primary purpose of this study is to provide treatment to patients who have participated on a prior protocol investigating Tanespimycin (KOS-953,17-AAG)

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Participated in and completed a previous Tanespimycin protocol without evidence of unacceptable toxicity and is deemed by the Investigator to be deriving benefit from the Tanespimycin drug as defined in the previous protocol
* All patients must rollover to this continuation protocol within 30 days of the last dose of Tanespimycin in the previous protocol, unless previously approved by the Medical Monitor
* All Adverse Events from the prior protocol, must have resolved to NCI CTCAE (v. 3.0) Grade <= 2
* The following laboratory results, within 10 days of Tanespimycin administration:
* Hemoglobin >= 8 g/dL
* Absolute neutrophils count >= 1.0x 10*9* /L
* Platelet count >= 50 x 10*9* /L
* Serum bilirubin <= 2 x ULN
* AST <= 2.5 ULN
* Serum creatinine <= 2 x ULN
* ECOG performance status of 0, 1 or 2
* Signed informed consent

Exclusion Criteria:

* Pre-existing neuropathy of CTCAE Grade >= 3 due to any cause
* Documented hypersensitivity reaction of CTCAE Grade >= 3 to prior therapy containing Cremophor (for those patients receiving Tanespimycin Injection)
* Pregnant or breast-feeding women
* Administration of chemotherapy, biological, immunotherapy or investigational agent (therapeutic or diagnostic), excluding Tanespimycin within 21 days prior to receipt of study medication
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-07; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
There is no Primary Outcome | No formal analysis of efficacy will occur

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx